CLINICAL TRIAL: NCT01267656
Title: Study to Evaluate the Product Feasibility of a Contact Lens Lubricating and Rewetting Drop
Brief Title: Study to Evaluate a Contact Lens Lubricating and Rewetting Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 684E
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye
Keywords: rewetting; lubricating; eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubricating and Rewetting Drops (Experimental): Lubricating and Rewetting Drops, after one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week.
  Interventions: Device: Lubricating and Rewetting Drops
- AMO Blink Contacts Lubricant Eye Drops (Active Comparator): AMO Blink Contacts Lubricant Eye Drops, After one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week
  Interventions: Device: AMO Blink Contacts Lubricant Eye Drops

INTERVENTIONS:
Device: Lubricating and Rewetting Drops — Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
  Arms: Lubricating and Rewetting Drops
Device: AMO Blink Contacts Lubricant Eye Drops — Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
  Arms: AMO Blink Contacts Lubricant Eye Drops

SUMMARY:
The objective of this study is to evaluate the product performance of investigational lubricating and rewetting drops.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Use a lens care system on a regular basis.
* Wear their habitual lenses (or be willing to wear lenses) a minimum of 8 hours per day.
* Willing to use drops 4 times per day.

Exclusion Criteria:

* Participating in a conflicting study.
* An active ocular disease, any corneal infiltrative response, or are using any ocular medications.
* Any scar or neovascularization within the central 4mm of the cornea.
* Any grade 2 or greater finding during the slit lamp examination
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* Aphakic.
* Amblyopic.
* Allergic to any component in the study care products.
* Have had any corneal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Su, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 168 participants enrolled and 166 participants treated. The study was a cross-over study, so the 166 participants received both treatment groups.
Groups:
- Lubricating and Rewetting Drops Then AMO Blink Contacts Lubric: Lubricating and Rewetting Drops, after one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week.
  Lubricating and Rewetting Drops: Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
  AMO Blink Contacts Lubricant Eye Drops, After one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week AMO Blink Contacts Lubricant Eye Drops: Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
- AMO Blink Contacts Lubricant Eye Drops Then Lubricating and Re: AMO Blink Contacts Lubricant Eye Drops, After one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week
  AMO Blink Contacts Lubricant Eye Drops: Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
  Lubricating and Rewetting Drops, after one week of using the first rewetting drops, the subjects will return for an exam and crossover to the second rewetting drops for one week.
  Lubricating and Rewetting Drops: Instill 1-2 rewetting drops in each eye at least QID (4 times per day) for one week.
Period: Overall Study
Arm/Group | Lubricating and Rewetting Drops Then AMO Blink Contacts Lubric | AMO Blink Contacts Lubricant Eye Drops Then Lubricating and Re
Started | 83 | 83
Completed | 82 | 82
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated participants were included in the analysis population.
Groups:
- Overall: The study was a cross-over study, so the 166 treated participants received both treatment groups.
Arm/Group | Overall
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Graded Slit Lamp Findings Greater Than Grade 2.
Description: Slit lamp findings for epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded 0 to 4, with 0 = none to 4 = severe. The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: At 1 week follow up
Population: There were 330 eyes evaluable for slit lamp findings in each group.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Lubricating and Rewetting Drops | AMO Blink Contacts Lubricant Eye Drops
Number analyzed (Participants) | 165 | 165
Number analyzed (eyes) | 330 | 330
eyes | 1 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were not coded. Therefore source vocabulary is not applicable.
Arm/Group | Lubricating and Rewetting Drops | AMO Blink Contacts Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/166
Other Adverse Events (participants affected / at risk) | 0/166 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.